CLINICAL TRIAL: NCT06214650
Title: Efficacy of a Combined Treatment With Abdominal Exercise and Radiofrequency in Postpartum Women With Diastasis Recti Abdominis
Brief Title: Diastasis Recti Abdominis and a Combined Treatment With Abdominal Exercise and Radiofrequency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, LOURDES PEÑA ROMERO, Principal Investigator, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lpena1
Record Dates: First submitted 2023-12-27; First posted 2024-01-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diastasis; Diastasis Recti; Diastasis Recti and Weakness of the Linea Alba; Diastasis Recti Abdominis
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency group (Experimental): All participants will be receive two interventions:
  1. A weekly session for 10 weeks with radiofrequency. It will be use the protocol of INDIBA. Each session will last 30 minutes.
  2. Participants will do an homely exercise protocol. This protocol will practise for 3 days at week.
  Interventions: Other: Radiofrequency
- Control group (Active Comparator): All participants will be receive two interventions:
  1. A weekly session for 10 weeks with radiofrequency. It will be use INDIBA without intensity such as a placebo. Each session will last 30 minutes.
  2. Participants will do an homely exercise protocol. This protocol will practise for 3 days at week.
  Interventions: Other: Control

INTERVENTIONS:
Other: Radiofrequency — Experimental group will receive the common exercise program associated with a radiofrequency treatment using INDIBA® (INDIBA Activ 7, Barcelona, INDIBA S.A.) at a frequency of 448 hertz. It will use the capacitive electrode as a method of preparation and vascularization of the superficial tissues and immediately, within the same session, the resistive electrode to stimulate deep tissues. This treatment is based on the protocols established by INDIBA® S.A.
  It will consist of one weekly diathermy session of thirty minutes during ten weeks. The use of diathermy will not be interrupted throughout the session.
  The common exercise program consist in a ten abdominal exercises (including recti abdominis, transversus and obliques). It will practised at home only just three days at week.
  Arms: Radiofrequency group
Other: Control — Control group will receive a weekly INDIBA® session in the abdominal area with the same protocol as the experimental group in athermic mode (placebo treatment) and the common exercise program. The session will last thirty minutes and will be carried out by the research physiotherapist during ten weeks.
  Arms: Control group

SUMMARY:
Diastasis recti abdominis is a pathology that appears in a high percentage of women during the postpartum period. However, there is little evidence about its treatment. The present protocol aims to evaluate the efficacy of radiofrequency as an alternative for the treatment of abdominal diastasis along with abdominal exercises compared to the only intervention through abdominal exercise.

An aleatory clinical testing will be conducted where 44 women diagnosed with diastasis recti abdominis in the postpartum period will be recruited. A common exercise protocol will be applied for two groups of participants, and both of them will have to be able to carry out the activities autonomously at home. In addition, control sessions will be held weekly for both groups where one of the groups, the control group (n=22), will receive radiofrequency therapy with the machine in athermic mode, while the other group, the experimental group (n=22), will receive a weekly session under the established diathermy protocol. The sessions will last 30 minutes and will take place for 10 consecutive weeks.

Three variables will be evaluated: the width of the diastasis measured in centimeters, life quality measured using the Short form (36) questionnaire, and the perception of the pain measured with the visual analogue scale. Three evaluations will be done: at the beginning of the study, after ten weeks and three months later.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with diastasis recti abdominis (DRA)
* Age range18-45 years old
* Women not DRA treated previously
* Women not diagnosed with umbilical hernia

Exclusion Criteria:

* DRA width less than 2.5cm
* Women diagnosed with intestinal disease such as irritable bowel syndrome (IBS) or Chron disease.
* Women looking for a new pregnancy or pregnant women.
* Women who can not receive diathermy treatment (e.g tumoral process, open wound in the abdominal area or any diathermy contraindication).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Width of the diastasis recti abdominis | It will be collected two measures to compare the changes: at baseline to the study and ten weeks later.
  The inter-recti diastasis will be measured with a transabdominal ultrasound using a lineal transductor. It will be assessed three measures: 2cm and 5cm above the umbilicus and 2cm below the umbilicus.

SECONDARY OUTCOMES:
Participant's quality of life | At baseline pre intervention and inmediately after the intervention (10 weeks later)
  Quality of life will be assessed using the Short form (36) questionnaire, which consist in thirty six questions about how pathology affects the participant's life.
Low back pain | At baseline pre intervention and inmediately after the intervention (10 weeks later)
  It will analysed the low back pain in the participants using the visual analogic scale (VAS). The participants will choose a level of pain (0-5) in the scale.